CLINICAL TRIAL: NCT01525836
Title: Recombinant Human Thrombopoietin in Combination With Rituximab Versus Low-dose Rituximab for the Treatment of Refractory ITP.
Brief Title: rhTPO Combining Rituximab Versus Low-dose Rituximab in Management of ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shandong Provincial Hospital (Other Government); Shenzhen Second People's Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-004
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-05

CONDITIONS: Purpura; Idiopathic Thrombocytopenic Purpura
Keywords: Purpura; Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination treatment group (Experimental): 120 enrolled patients are randomly picked up to take Rituximab in combination with Rh-TPO at the indicated dose.
  Interventions: Drug: rituximab; recombinant human thrombopoietin (rhTPO)
- single treatment group (Active Comparator): 120 enrolled patients are randomly picked up to take Rituximab at the indicated dose.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: rituximab; recombinant human thrombopoietin (rhTPO) — patients in recombination treatment group take Rituximab( intravenously ,100 mg weekly for 4 consecutive weeks); in combination with Rh-TPO( subcutaneously , 300U/kg for 14 consecutive days,followed by flexible treating dosage so as to keep the platelet count above 50×10^9/L until the 29th day)
  Other Names: Recombinant Human Thrombopoietin; Recombinant Human TPO; rhTPO combine with Rituximab; Recombinant Human Thrombopoietin combine with Rituximab; Recombinant Human TPO combine with Rituximab
  Arms: combination treatment group
Drug: Rituximab — patients in recombinant treatment group take Rituximab intravenously at 100 mg weekly for 4 consecutive weeks（Day 1,8,15,22)
  Arms: single treatment group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 13 well-known hospitals in China. In order to report the efficacy and safety of Recombinant Human thrombopoietin combining with Rituximab for the treatment of adults with refractory immune thrombocytopenia (ITP), compared to conventional Rituximab therapy.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 240 refractory ITP adult patients from 14 medical centers in China. One part of the participants are randomly selected to receive recombinant human thrombopoietin (given subcutaneously at a dose of 300 Units/kg for 14 consecutive days,following with a flexible dosage depending on platelet count until the 29th day), combining with rituximab (given intravenously at a dose of 100 mg weekly for 4 weeks, i.e. Day 1, 8, 15, 22; the others are selected to receive low-dose of rituximab treatment (given intravenously at a dose of 100 mg weekly, i.e. Day 1, 8, 15, 22). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of the combination therapy compared to conventional rituximab therapy for the treatment of adults with refractory ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.
5. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received high-dose steroids or [2] intravenous immunoglobulin transfusion(IVIG)in the 3 weeks prior to the start of the study.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections. Severe medical condition (lung, hepatic or renal disorder) other than ITP. 4.Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)

5.Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.

6.Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.

7.Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 3 months per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L
Evaluation of platelet response (Response) | The time frame is up to 3 months per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia.
Evaluation of platelet response (No Response) | The time frame is up to 3 months per subject
  NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
Evaluation of platelet response (relapses) | The time frame is up to 3 months per subject
  A relapses was defined as platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

SECONDARY OUTCOMES:
The number and frequency of therapy associated adverse events | up to 3 months per subject

CONTACTS AND LOCATIONS:
Overall Officials: Minf Hou, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Medeot M, Zaja F, Vianelli N, Battista M, Baccarani M, Patriarca F, Soldano F, Isola M, De Luca S, Fanin R. Rituximab therapy in adult patients with relapsed or refractory immune thrombocytopenic purpura: long-term follow-up results. Eur J Haematol. 2008 Sep;81(3):165-9. doi: 10.1111/j.1600-0609.2008.01100.x. Epub 2008 May 27. PMID 18510702
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Background] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333
- [Derived] Zhou H, Xu M, Qin P, Zhang HY, Yuan CL, Zhao HG, Cui ZG, Meng YS, Wang L, Zhou F, Wang X, Li DQ, Bi KH, Zhu CS, Guo CS, Chu XX, Wu QC, Liu XG, Dong XY, Li J, Peng J, Hou M. A multicenter randomized open-label study of rituximab plus rhTPO vs rituximab in corticosteroid-resistant or relapsed ITP. Blood. 2015 Mar 5;125(10):1541-7. doi: 10.1182/blood-2014-06-581868. Epub 2015 Jan 9. PMID 25575541